CLINICAL TRIAL: NCT02348723
Title: Randomized Evaluation of Dabigatran Etexilate Compared to warfarIn in pulmonaRy Vein Ablation: Assessment of an Uninterrupted periproCedUral alntIcoagulation sTrategy (The RE-CIRCUIT Trial)
Brief Title: Uninterrupted Dabigatran Etexilate in Comparison to Uninterrupted Warfarin in Pulmonary Vein Ablation (RE-CIRCUIT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.204; 2014-003890-40 (EudraCT Number)
Record Dates: First submitted 2015-01-27; First posted 2015-01-28 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; Dabigatran

ARMS (2):
- Dabigatran Etexilate 150mg (Experimental): Patients receiving Dabigatran Etexilate 150mg twice daily dosing (BID)
  Interventions: Drug: Dabigatran Etexilate 150mg
- Warfarin (Active Comparator): Patients receiving Warfarin to keep International Normalized Ratio (INR) between 2.0 - 3.0
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin — Patients receiving Warfarin to keep International Normalized Ratio (INR)between 2.0 - 3.0
  Arms: Warfarin
Drug: Dabigatran Etexilate 150mg — Patients receiving Dabigatran Etexilate 150mg twice daily dosing (BID)
  Arms: Dabigatran Etexilate 150mg

SUMMARY:
The primary objective of this trial is to assess the safety of an uninterrupted dabigatran etexilate periprocedural anticoagulant regimen compared to an uninterrupted warfarin regimen in Non-Valvular Atrial Fibrillation (NVAF) patients undergoing Atrial Fibrillation (AF) ablation in a PROBE (Prospective, randomized, open label, blinded end point) active controlled study.

Secondary objectives are to assess additional safety endpoints and efficacy in this clinical setting.

It is not intended to assess confirmatory hypothesis, this is an exploratory study.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients aged >= 18 years.
* Patients eligible for treatment with dabigatran etexilate 150 mg b.i.d. according to local label.
* Treatment naïve patients or patients on oral anticoagulant treatment with a Vitamin K Antagonist (VKA), dabigatran etexilate, rivaroxaban, apixaban or edoxaban.
* Patient with paroxysmal or persistent NVAF with a planned catheter ablation for AF unless it is performed an investigational ablation technique.
* AF must have been documented at least once either by ECG, Holter monitoring, loop recorder, telemetry, trans-telephonic monitoring, pacemaker or cardiac defibrillator read outs within 24 months prior to screening (Visit 1).
* The patient must be able to give informed consent in accordance with International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) guidelines and local legislation and/or regulations.

Exclusion criteria:

* Patients with permanent AF.
* Patients with AF felt to be secondary to an obvious reversible cause such as, but not limited to, an acute myocardial infarction, pulmonary embolism, recent surgery, pericarditis or thyrotoxicosis.
* Patients with Left Atrium (LA) size >= 60 mm
* Patients with contraindications to systemic anticoagulation with heparin, warfarin or dabigatran etexilate
* Patients with a known allergy to warfarin tablets and it excipients or to dabigatran etexilate or its excipients
* Mechanical or biological heart valve prosthesis
* Severe renal impairment (estimated Creatinine Clearance (CrCl) calculated by Cockcroft-Gault equation) <30mL/min at screening
* Stroke within 1 month prior to screening visit
* Major surgery per investigator judgement within the previous month prior to screening.
* Patient has received an organ transplant or is on a waiting list for an organ transplant
* History of intracranial haemorrhage, intraocular, spinal, retroperitoneal or non-traumatic intra-articular bleeding
* Gastrointestinal haemorrhage within one month prior to screening, unless, in the opinion of the investigator, the cause has been permanently eliminated (e.g. by surgery).
* Major bleeding episode (ISTH definition) one month prior to the screening visit.
* Haemorrhagic disorder or bleeding diathesis (e.g. von Willebrand disease, haemophilia A or B or other hereditary bleeding disorder, history of spontaneous intra-articular bleeding, history of prolonged bleeding after surgery/intervention)
* Anaemia (haemoglobin <10g/dL) or thrombocytopenia including heparin-induced thrombocytopenia (platelet count <100 x 10^9/L) at screening
* Recent malignancy or radiation therapy (<=6 months prior to screening) unless, in the opinion of the Investigator, the estimated life expectancy is greater than 36 months
* Active liver disease as indicated by at least one of the following:

  -- Prior and persistent alanine aminotransferase or Aspartate transaminase or alkaline phosphatase >3x upper limit of normal and/or -- Known active hepatitis C and/or -- Known active hepatitis B and/or -- Known active hepatitis A
* Need for continued treatment with systemic ketoconazole, itraconazole, posaconazole, cyclosporine, tacrolimus, dronedarone, rifampicin, phenytoin, carbamazepine, St. John's Wort or any cytotoxic/myelosuppressive therapy.
* Pre-menopausal (last menstruation <=1 year prior to screening) who:

  * Are pregnant or breast-feeding or plan to become pregnant during study or
  * Are not surgically sterile or
  * Are of child bearing potential and not practising two acceptable method of birth control, or do not plan to continue practising an acceptable method of birth control throughout the trial
* Patients who have participated in another trial with an investigational drug or device within the past 30 days preceding the screening visit or are participating in another trial (patients participating in an observational study only will not be excluded)
* Patients not willing or able to comply with the protocol requirements or considered unreliable by the Investigator concerning the requirements for follow-up during the study and/or compliance with study drug administration, who have a life expectancy less than the expected duration of the trial due to concomitant disease and/or subjects who are institutionalised due to official or court orders and/or vulnerable subjects who are dependent on the Sponsor or the Investigator or the site, or patients who have any condition which in the opinion of the Investigator, would not allow safe participation in the study (e.g. drug addiction, alcohol abuse).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (87):
- United States (21):
  - Arkansas Cardiology, PA, Little Rock, Arkansas
  - Mission Cardiovascular Research Institute, Fremont, California
  - University of California, Sacramento, California
  - Mercy Medical Group, a service of Dignity Health Medical Foundation, Sacramento, California
  - University of California, San Francisco, California
  - Southwest Florida Research, LLC, Naples, Florida
  - University of South Florida, Tampa, Florida
  - Elkhart General Healthcare System, Elkhart, Indiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - New York Methodist Hospital, Brooklyn, New York
  - University at Buffalo, The State University of New York, Buffalo, New York
  - Staten Island University Hospital, Staten Island, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Tennessee Methodist Physicians, Memphis, Tennessee
  - North Texas Heart Center, Dallas, Texas
  - St Luke's Health Baylor College of Medicine Med Center, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Providence Regional Medical Center, Everett, Washington
- Belgium (6):
  - Bonheiden - HOSP Imelda, Bonheiden
  - Brussels - UNIV UZ Brussel, Brussels
  - UNIV UZ Gent, Ghent
  - Centre Hospitalier Universitaire de Liège, Liège
  - Antwerpen - HOSP ZNA Middelheim - Pneumo, Middelheim
  - Brussels - HOSP Europe (Ste-Elisabeth), Uccle
- Canada (6):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Victoria Cardiac Arrhythmia Trials Inc., Victoria, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - CHUS Fleurimont, Sherbrooke, Quebec
  - IUCPQ (Laval University), Québec
- France (7):
  - HOP Nord Michallon, La Tronche
  - HOP Timone, Marseille
  - CLI Nouvelles Cliniques Nantaises,Cardio,Nantes Cedex 2, Nantes
  - HOP Salpêtrière, Cardio, Paris, Paris
  - HOP Européen G. Pompidou, Paris
  - HOP Haut-Lévêque, Pessac
  - HOP CHU Nancy Brabois, Cardiologie, Vandœuvre-lès-Nancy
- Germany (7):
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Ulm, Ulm
- Italy (6):
  - Ospedale Generale Regionale "Miulli", Acquaviva Delle Fonti (BA)
  - A.S.O.S. Croce e Carle, Cuneo
  - Osp.dell'Angelo, Mestre-Venezia
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Centro Cardiologico Monzino-IRCCS, Milan
  - Policlinico Casilino U.O. Cardiologia, Roma
- Japan (10):
  - Anjo-kosei Hospital, Aichi, Anjo
  - Nagoya City East Medical Center, Aichi, Nagoya
  - Nagoya University Hospital, Aichi, Nagoya
  - Japanese Red Cross Nagoya Daini Hospital, Aichi, Nagoya
  - Hirosaki University Hospital, Aomori, Hirosaki
  - New Tokyo Heart Clinic, Chiba, Matsudo
  - Shonan Kamakura General Hospital, Kanagawa, Kamakura
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Nippon Medical School Hospital, Tokyo, Bunkyo-Ku
  - Tokyo Medical University Hachioji Medical Center, Tokyo, Hachioji
- Netherlands (5):
  - VU Medisch Centrum, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Radboud Universitair Medisch Centrum, Nijmegen
- Russia (6):
  - Heart&Vessels Diseases,Cardiol&Cardiovas.SurgeryDep,Kamerovo, Kemerovo
  - Instit.of Surgery na Vishnevskiy,Treatm.of comp.arrhythm.dep, Moscow
  - North-Westrn Fed.med.res.cntr,Almazov Interven.arrhythmo.dep, Saint Petersburg
  - City Pokrovskiy Hospital, Cardiology Dept., Saint Petersburg, Saint Petersburg
  - Tyumen Cardiology Center, Dept.of Cardiac Arrhythmia, Tyumen
  - Yaroslavl Regional Clin. Hospital, Dept. Endocrinology, Yaroslavl
- Spain (4):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital La Paz, Madrid
  - Hospital Virgen del Rocío, Seville
  - Hospital Álvaro Cunqueiro, Vigo (Pontevedra)
- United Kingdom (9):
  - Royal Bournemouth and Christchurch Hospital, Bournemouth
  - Royal Sussex County Hospital, Brighton
  - Papworth Hospital, Cambridge
  - Golden Jubilee National Hospital, Clydebank, Clydebank
  - Castle Hill Hopsital, Cottingham
  - Leeds General Infirmary, Leeds
  - St Bartholomew's Hospital, London
  - James Cook University Hospital, Middlesbrough
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Kimata A, Nogami A, Yamasaki H, Ohigashi T, Gosho M, Igarashi M, Sekiguchi Y, Ieda M, Calkins H, Aonuma K. Optimal interruption time of dabigatran oral administration to ablation (O-A time) in patients with atrial fibrillation: Integrated analysis of 2 randomized controlled clinical trials. J Cardiol. 2021 Jun;77(6):652-659. doi: 10.1016/j.jjcc.2020.12.010. Epub 2021 Jan 25. PMID 33509678
- [Derived] Hohnloser SH, Calkins H, Willems S, Verma A, Schilling R, Okumura K, Nordaby M, Kleine E, Biss B, Gerstenfeld EP; RE-CIRCUIT(R) investigators. Regional differences in patient characteristics and outcomes during uninterrupted anticoagulation with dabigatran versus warfarin in catheter ablation of atrial fibrillation: the RE-CIRCUIT study. J Interv Card Electrophysiol. 2019 Aug;55(2):145-152. doi: 10.1007/s10840-019-00518-x. Epub 2019 Feb 13. PMID 30758702
- [Derived] Calkins H, Willems S, Gerstenfeld EP, Verma A, Schilling R, Hohnloser SH, Okumura K, Serota H, Nordaby M, Guiver K, Biss B, Brouwer MA, Grimaldi M; RE-CIRCUIT Investigators. Uninterrupted Dabigatran versus Warfarin for Ablation in Atrial Fibrillation. N Engl J Med. 2017 Apr 27;376(17):1627-1636. doi: 10.1056/NEJMoa1701005. Epub 2017 Mar 19. PMID 28317415

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomly assigned to dabigatran etexilate 150 mg twice daily or warfarin in a 1:1 ratio and remained on this treatment for the duration of the trial. 678 subjects were randomised and 676 were treated.
Groups:
- Dabigatran Etexilate 150 mg: Patients receiving Dabigatran Etexilate 150 mg capsule orally twice daily (BID);
  1 capsule 150 mg twice daily (total daily dose 300 mg)
- Warfarin: Patients receiving Warfarin tablet orally;
  1, 3, and 5 mg (dose adjusted to International normalized ratio (INR) target range)
Period: Overall Study
Arm/Group | Dabigatran Etexilate 150 mg | Warfarin
Started | 338 | 338
Completed | 310 | 312
Not Completed | 28 | 26
Not completed — No ablation | 21 | 20
Not completed — Non-compliant with Protocol | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Consent withdrawn | 1 | 3
Not completed — Reason other than specified | 1 | 1
Not completed — Adverse Event | 3 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set (TS) included all patients who were randomised and subsequently treated with at least 1 tablet/capsule.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate 150 mg | Warfarin | Total
Number analyzed (Participants) | 338 | 338 | 676
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (10.33) | 59.4 (10.29) | 59.3 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 81 | 174
  Male | 245 | 257 | 502

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Major Bleeding Events (MBEs), as Defined by the International Society on Thrombosis and Haemostasis (ISTH)
Description: Major bleeds were defined according to the ISTH definition of a major bleed, as follows
  * Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome and/or
  * Bleeding associated with a reduction in haemoglobin of at least 2 g/dL (1.24 mmol/L), or leading to transfusion of 2 or more units of blood or packed cells. and/or
  * Fatal bleed
  These are based on adjudicated data (blinded evaluation)
  Point estimates for the incidence of ISTH MBEs and their 2-sided 95% confidence intervals (CI), based on the normal approximation of independent binomial distribution without stratification, are presented.
Time Frame: during and up to 2 months post-ablation
Population: The ablation set (AS) was the primary analysis set and included all patients in the treated set (TS) who started the ablation procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dabigatran Etexilate 150 mg | Warfarin
Number analyzed (Participants) | 317 | 318
percentage of participants | 1.6 [0.2 to 2.9] | 6.9 [4.1 to 9.7]
Statistical Analysis 1: Comparison: Dabigatran Etexilate 150 mg vs Warfarin; The risk difference between dabigatran etexilate vs. warfarin, its 2-sided 95% CI, and corresponding p-value are presented; Test type: Superiority or Other; p = 0.0009, Chi-squared; Risk Difference (RD) % = -5.3, 95% CI 2-sided [-8.4 to -2.2]

2. Secondary Outcome: Incidence of the Composite of Stroke, Systemic Embolism, or Transient Ischemic Attack (TIA)
Description: Stroke was defined as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of haemorrhage or infarction.
  Systemic embolism was defined as an acute vascular occlusion of the extremities or any organ (kidneys, mesenteric arteries, spleen, retina or grafts) and was to be documented by angiography, surgery, scintigraphy or autopsy.
  Transient ischemic attack was defined as a transient episode of focal neurological dysfunction caused by brain, spinal cord, or retinal ischemia, without acute infarction.
  These are based on adjudicated data (blinded evaluation).
  Percentage of patients with composite of stroke, systemic embolism, or transient ischemic attack (TIA) is presented
Time Frame: during and up to 2 months post-ablation
Population: AS
Measure: Number; unit: percentage of participants
Arm/Group | Dabigatran Etexilate 150 mg | Warfarin
Number analyzed (Participants) | 317 | 318
percentage of participants | 0.0 | 0.3

3. Secondary Outcome: Incidence of Minor Bleeding Events
Description: Minor bleeds were clinical bleeds that did not fulfil the criteria for major bleeds. Percentage of patients with Minor bleeding events are presented.
  These are based on adjudicated data (blinded evaluation)
Time Frame: during and up to 2 months post-ablation
Population: AS
Measure: Number; unit: percentage of participants
Arm/Group | Dabigatran Etexilate 150 mg | Warfarin
Number analyzed (Participants) | 317 | 318
percentage of participants | 18.6 | 17.0

4. Secondary Outcome: Incidence of ISTH MBE, Stroke, Systemic Embolism, or TIA (Composite Endpoint Combining Safety and Efficacy
Description: Percentage of patients with ISTH MBE, stroke, systemic embolism, or TIA (composite endpoint combining safety and efficacy) are presented.
  These are based on adjudicated data (blinded evaluation)
Time Frame: during and up to 2 months post-ablation
Population: AS
Measure: Number; unit: percentage of participants
Arm/Group | Dabigatran Etexilate 150 mg | Warfarin
Number analyzed (Participants) | 317 | 318
percentage of participants | 1.6 | 7.2

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) which occurred after the first dose of trial medication up to 6 days after the last dose of trial medication; up to 225 days
Arm/Group | Dabigatran Etexilate 150 mg | Warfarin
Serious Adverse Events (participants affected / at risk) | 63/338 | 75/338
Other Adverse Events (participants affected / at risk) | 68/338 | 65/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 150 mg (N=338) | Warfarin (N=338)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 13
Atrial flutter (Cardiac disorders) | 20 | 19
Atrial tachycardia (Cardiac disorders) | 2 | 1
Atrial thrombosis (Cardiac disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 4
Coronary artery disease (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 2 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 3
Malaise (General disorders) | 0 | 1
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 4
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 | 1
Bleeding time prolonged (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1
Peripheral nerve paresis (Nervous system disorders) | 0 | 1
Phrenic nerve paralysis (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 6
Haemorrhage (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 150 mg (N=338) | Warfarin (N=338)
Atrial fibrillation (Cardiac disorders) | 40 | 38
Palpitations (Cardiac disorders) | 16 | 19
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.